CLINICAL TRIAL: NCT06640829
Title: Added Sugar Intake and Brain Structure and Function
Acronym: GAINS BRAINS
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Collaborators: Center for Children's Healthy Lifestyles & Nutrition (Unknown)
Responsible Party: Sponsor
Other Study IDs: STUDY00149236
Record Dates: First submitted 2024-08-29; First posted 2024-10-15 (Actual); Results first posted 2025-07-04 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-06

CONDITIONS: Child Development
Keywords: Added sugars; Dietary intake; Brain health; Child development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ADORE GAINS Participants: Children's who participated in the ADORE GAINS study were invited to participate as their body composition and dietary intake was collected during their infancy and toddlerhood.

SUMMARY:
The purpose of this study is to learn if there is a relationship between added sugar intake during pregnancy, infancy, and toddlerhood and the brain's structure and function at 5-6 years old.

ELIGIBILITY:
Inclusion Criteria:

* Participated in the ADORE GAINS study (R01 DK118220).
* Age at participation 5-6 years old.

Exclusion Criteria:

* Did not participated in the ADORE GAINS study.
* Younger than 5 and older than 6.
* Autism diagnosis

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants received an invitation to participate in this study if they were enrolled in the ADORE GAINS study as an infant and toddler.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2023-03-23 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Holly Hull, PhD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ADORE GAINS Participants
Started | 42
Completed | 40
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: 42 participants enrolled, two participants did not complete the study
Arm/Group | ADORE GAINS Participants
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 5.77 (0.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 28
  More than one race | 6
  Unknown or Not Reported | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 19
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Percent of energy (kilocalories) from added sugars at age 5-6 years [Mean (Standard Deviation); unit: Percentage of kilocalorie intake] — Population: two participants had incomplete/invalid dietary data
  Percentage of kilocalorie intake
    number analyzed (Participants) | 40
    (all) | 13.89 (5.52)
Percent of energy (kilocalories) from fructose at age 5-6 years [Mean (Standard Deviation); unit: Percentage of kilocalorie intake] — Population: two participants had incomplete/invalid dietary data
  Percentage of kilocalorie intake
    number analyzed (Participants) | 40
    (all) | 4.68 (2.05)

OUTCOME MEASURES:

1. Primary Outcome: Added Sugars Intake Relationship to Brain Structure
Description: Assess the impact of added sugars intake measured by 24-hour dietary intake on brain structure, quantified as brain volume, via an MRI 3D MPRAGE and fMRI sequencing. Maternal dietary intake information was collected at baseline in the ADORE study between 12-20 weeks gestation. Offspring dietary intake information was collected at 6-months, 12-months, and 24-months of age in the ADORE GAINS study. Dietary intake, MRI, EEG, and cognition were assessed at age 5-6 years in the present study.
Time Frame: Day 1 in the present study (age 5-6 years old); Baseline, 6 months, 12 months and 24 months in the ADORE GAINS study; Baseline (12-20 weeks gestation) in the ADORE study;
Population: only 13 participants had complete/valid dietary data and usable MRI data
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | ADORE GAINS Participants
Number analyzed (Participants) | 13
Pearson correlation coefficient
  Left Hippocampal Volume and Percent of Calories from Added Sugars at age 5-6 years | 0.119
  Right Hippocampal Volume and Percent of Calories from Added Sugars at age 5-6 years | -0.231
  Left Hippocampal Volume and Percent of Calories from Added Sugars at age 6 months | 0.345
  Right Hippocampal Volume and Percent of Calories from Added Sugars at age 6 months | 0.384
  Left Hippocampal Volume and Percent of Calories from Added Sugars at age 12 months | 0.176
  Right Hippocampal Volume and Percent of Calories from Added Sugars at age 12 months | -0.202
  Left Hippocampal Volume and Percent of Calories from Added Sugars at age 24 months | 0.242
  Right Hippocampal Volume and Percent of Calories from Added Sugars at age 24 months | 0.016
  Left Hippocampal Volume and Maternal Prenatal Percent of Calories from Added Sugars | -0.045
  Right Hippocampal Volume and Maternal Prenatal Percent of Calories from Added Sugars | -0.502

2. Primary Outcome: Added Sugars Intake Relationship to Brain Function
Description: Assess the impact of added sugars intake measured by 24-hour dietary intake on the brain's function via EEG (task-based (Go/NoGo task) event-related potentials (ERPs)) to identify brain activity related to inhibitory control, quantified by amplitude for the Go and NoGo conditions. Maternal dietary intake information was collected at baseline in the ADORE study between 12-20 weeks gestation. Offspring dietary intake information was collected at 6-months, 12-months, and 24-months of age in the ADORE GAINS study. Dietary intake, MRI, EEG, and cognition were assessed at age 5-6 years in the present study.
Time Frame: as for outcome 1
Population: only 18 participants had both complete/valid dietary data and EEG data
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | ADORE GAINS Participants
Number analyzed (Participants) | 18
Pearson correlation coefficient
  Go Trials N2 Amplitude and Percent of Calories from Added Sugars at age 5-6 years | 0.059
  No-Go Trials N2 Amplitude and Percent of Calories from Added Sugars at age 5-6 years | -0.016
  Go Trials P3 Amplitude and Percent of Calories from Added Sugars at age 5-6 years | -0.045
  No-Go Trials P3 Amplitude and Percent of Calories from Added Sugars at age 5-6 years | 0.090
  Go Trials N2 Amplitude and Percent of Calories from Added Sugars at age 6 months | 0.481
  No-Go Trials N2 Amplitude and Percent of Calories from Added Sugars at age 6 months | 0.404
  Go Trials P3 Amplitude and Percent of Calories from Added Sugars at age 6 months | -0.183
  No-Go Trials P3 Amplitude and Percent of Calories from Added Sugars at age 6 months | -0.095
  Go Trials N2 Amplitude and Percent of Calories from Added Sugars at age 12 months | 0.534
  No-Go Trials N2 Amplitude and Percent of Calories from Added Sugars at age 12 months | 0.459
  Go Trials P3 Amplitude and Percent of Calories from Added Sugars at age 12 months | -0.358
  No-Go Trials P3 Amplitude and Percent of Calories from Added Sugars at age 12 months | -0.176
  Go Trials N2 Amplitude and Percent of Calories from Added Sugars at age 24 months | -0.083
  No-Go Trials N2 Amplitude and Percent of Calories from Added Sugars at age 24 months | -0.088
  Go Trials P3 Amplitude and Percent of Calories from Added Sugars at age 24 months | 0.028
  No-Go Trials P3 Amplitude and Percent of Calories from Added Sugars at age 24 months | -0.042
  Go Trials N2 Amplitude and Maternal Prenatal Percent of Calories from Added Sugars | 0.051
  No-Go Trials N2 Amplitude and Maternal Prenatal Percent of Calories from Added Sugars | 0.120
  Go Trials P3 Amplitude and Maternal Prenatal Percent of Calories from Added Sugars | -0.285
  No-Go Trials P3 Amplitude and Maternal Prenatal Percent of Calories from Added Sugars | -0.224

3. Primary Outcome: Fructose Intake Relationship to Brain Structure
Description: Assess the impact of fructose intake measured by 24-hour dietary intake on brain structure, quantified as brain volume, via an MRI 3D MPRAGE and fMRI sequencing. Maternal dietary intake information was collected at baseline in the ADORE study between 12-20 weeks gestation. Offspring dietary intake information was collected at 6-months, 12-months, and 24-months of age in the ADORE GAINS study. Dietary intake, MRI, EEG, and cognition were assessed at age 5-6 years in the present study.
Time Frame: as for outcome 1
Population: only 13 participants had complete/valid dietary data and usable MRI data
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | ADORE GAINS Participants
Number analyzed (Participants) | 13
Pearson correlation coefficient
  Left Hippocampal Volume and Percent of Calories from Fructose at age 5-6 years | -0.220
  Right Hippocampal Volume and Percent of Calories from Fructose at age 5-6 years | -0.413
  Left Hippocampal Volume and Percent of Calories from Fructose at age 6 months | -0.730
  Right Hippocampal Volume and Percent of Calories from Fructose at age 6 months | -0.071
  Left Hippocampal Volume and Percent of Calories from Fructose at age 12 months | 0.132
  Right Hippocampal Volume and Percent of Calories from Fructose at age 12 months | -0.535
  Left Hippocampal Volume and Percent of Calories from Fructose at age 24 months | -0.389
  Right Hippocampal Volume and Percent of Calories from Fructose at age 24 months | -0.213
  Left Hippocampal Volume and Maternal Prenatal Percent of Calories from Fructose | -0.252
  Right Hippocampal Volume and Maternal Prenatal Percent of Calories from Fructose | -0.466

4. Primary Outcome: Fructose Intake Relationship to Brain Function
Description: Assess the impact of fructose intake measured by 24-hour dietary intake on the brain's function via EEG (task-based (Go/NoGo task) event-related potentials (ERPs)) to identify brain activity related to inhibitory control, quantified by amplitude for the Go and NoGo conditions. Maternal dietary intake information was collected at baseline in the ADORE study between 12-20 weeks gestation. Offspring dietary intake information was collected at 6-months, 12-months, and 24-months of age in the ADORE GAINS study. Dietary intake, MRI, EEG, and cognition were assessed at age 5-6 years in the present study.
Time Frame: as for outcome 1
Population: only 18 participants had both complete/valid dietary data and EEG data
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | ADORE GAINS Participants
Number analyzed (Participants) | 18
Pearson correlation coefficient
  Go Trials N2 Amplitude and Percent of Calories from Fructose at age 5-6 years | -0.014
  No-Go Trials N2 Amplitude and Percent of Calories from Fructose at age 5-6 years | 0.018
  Go Trials P3 Amplitude and Percent of Calories from Fructose at age 5-6 years | -0.129
  No-Go Trials P3 Amplitude and Percent of Calories from Fructose at age 5-6 years | -0.275
  Go Trials N2 Amplitude and Percent of Calories from Fructose at age 6 months | -0.555
  No-Go Trials N2 Amplitude and Percent of Calories from Fructose at age 6 months | -0.331
  Go Trials P3 Amplitude and Percent of Calories from Fructose at age 6 months | 0.355
  No-Go Trials P3 Amplitude and Percent of Calories from Fructose at age 6 months | 0.416
  Go Trials N2 Amplitude and Percent of Calories from Fructose at age 12 months | 0.057
  No-Go Trials N2 Amplitude and Percent of Calories from Fructose at age 12 months | 0.152
  Go Trials P3 Amplitude and Percent of Calories from Fructose at age 12 months | 0.045
  No-Go Trials P3 Amplitude and Percent of Calories from Fructose at age 12 months | 0.040
  Go Trials N2 Amplitude and Percent of Calories from Fructose at age 24 months | -0.116
  No-Go Trials N2 Amplitude and Percent of Calories from Fructose at age 24 months | -0.110
  Go Trials P3 Amplitude and Percent of Calories from Fructose at age 24 months | 0.050
  No-Go Trials P3 Amplitude and Percent of Calories from Fructose at age 24 months | 0.076
  Go Trials N2 Amplitude and Maternal Prenatal Percent of Calories from Fructose | 0.414
  No-Go Trials N2 Amplitude and Maternal Prenatal Percent of Calories from Fructose | 0.507
  Go Trials P3 Amplitude and Maternal Prenatal Percent of Calories from Fructose | -0.463
  No-Go Trials P3 Amplitude and Maternal Prenatal Percent of Calories from Fructose | -0.600

5. Secondary Outcome: Added Sugars Intake Relationship to Cognition Specifically Attention Development
Description: Assess the impact of added sugars intake measured by 24-hour dietary intake on cognition via a Dimensional Change Card Sort (DCCS) task measuring attention development. Maternal dietary intake information was collected at baseline in the ADORE study between 12-20 weeks gestation. Offspring dietary intake information was collected at 6-months, 12-months, and 24-months of age in the ADORE GAINS study. Dietary intake, MRI, EEG, and cognition were assessed at age 5-6 years in the present study.
Time Frame: Day 7 in the present study (age 5-6 years old); Baseline, 6 months, 12 months and 24 months in the ADORE GAINS study; Baseline (12-20 weeks gestation) in the ADORE study;
Population: three participants either had incomplete/invalid dietary data and/or did not complete the cognitive test
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | ADORE GAINS Participants
Number analyzed (Participants) | 39
Pearson correlation coefficient
  DCCS Pre-Switch Score and Percent of Calories from Added Sugars at age 5-6 years | 0.163
  DCCS Post-Switch Score and Percent of Calories from Added Sugars at age 5-6 years | -0.076
  DCCS Borders Score and Percent of Calories from Added Sugars at age 5-6 years | -0.031
  DCCS Post-Switch Score and Percent of Calories from Added Sugars at age 6 months | -0.374
  DCCS Borders Score and Percent of Calories from Added Sugars at age 6 months | -0.259
  DCCS Pre-Switch Score and Percent of Calories from Added Sugars at age 12 months | 0.151
  DCCS Post-Switch Score and Percent of Calories from Added Sugars at age 12 months | 0.020
  DCCS Borders Score and Percent of Calories from Added Sugars at age 12 months | 0.037
  DCCS Pre-Switch Score and Percent of Calories from Added Sugars at age 24 months | 0.001
  DCCS Post-Switch Score and Percent of Calories from Added Sugars at age 24 months | -0.283
  DCCS Borders Score and Percent of Calories from Added Sugars at age 24 months | -0.108
  DCCS Pre-Switch Score and Maternal Prenatal Percent of Calories from Added Sugars | 0.171
  DCCS Post-Switch Score and Maternal Prenatal Percent of Calories from Added Sugars | -0.324
  DCCS Borders Score and Maternal Prenatal Percent of Calories from Added Sugars | -0.023

6. Secondary Outcome: Added Sugars Intake Relationship to Cognition Specifically Vocabulary Receptiveness
Description: Assess the impact of added sugars intake measured by 24-hour dietary intake on cognition via Peabody Picture Vocabulary Test measuring vocabulary receptiveness. Maternal dietary intake information was collected at baseline in the ADORE study between 12-20 weeks gestation. Offspring dietary intake information was collected at 6-months, 12-months, and 24-months of age in the ADORE GAINS study. Dietary intake, MRI, EEG, and cognition were assessed at age 5-6 years in the present study.
Time Frame: as for outcome 5
Population: three participants either had incomplete/invalid dietary data and/or did not complete the cognitive test
Measure: Number; unit: Pearson correlation coefficient
Arm/Group | ADORE GAINS Participants
Number analyzed (Participants) | 39
Pearson correlation coefficient
  PPVT Standard Score and Percent of Calories from Added Sugars at age 5-6 years | 0.118
  PPVT Percentile and Percent of Calories from Added Sugars at age 5-6 years | 0.124
  PPVT Standard Score and Percent of Calories from Added Sugars at age 6 months | 0.062
  PPVT Percentile and Percent of Calories from Added Sugars at age 6 months | 0.020
  PPVT Standard Score and Percent of Calories from Added Sugars at age 12 months | 0.035
  PPVT Percentile and Percent of Calories from Added Sugars at age 12 months | 0.043
  PPVT Standard Score and Percent of Calories from Added Sugars at age 24 months | -0.092
  PPVT Percentile and Percent of Calories from Added Sugars at age 24 months | -0.150
  PPVT Standard Score and Maternal Prenatal Percent of Calories from Added Sugars | -0.045
  PPVT Percentile and Maternal Prenatal Percent of Calories from Added Sugars | -0.126

ADVERSE EVENTS:
Time Frame: Collected for the duration of study visits, an average of 7 days
Arm/Group | ADORE GAINS Participants
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-19): https://cdn.clinicaltrials.gov/large-docs/29/NCT06640829/Prot_SAP_000.pdf